CLINICAL TRIAL: NCT03618225
Title: Duloxetine Role in Reducing Opioid Consumption After Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Assisstant professor of Anesthesia ICU and pain Relief, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORG0006563
Record Dates: First submitted 2018-07-14; First posted 2018-08-07 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Post-thoracotomy Pain
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- duloxetine group (Active Comparator): duloxetine 60 mg orally 2 hours before the surgical procedure and at 24 hours after the surgical procedure.
  Interventions: Drug: Oral Duloxetine 60mg
- placebo pill group (Placebo Comparator): placebo pill orally 2 hours before the surgical procedure and at 24 hours after the surgical procedure.
  Interventions: Drug: placebo pill

INTERVENTIONS:
Drug: Oral Duloxetine 60mg — duloxetine 60 mg orally 2 hours before the surgical procedure and at 24 hours after the surgical procedure
  Arms: duloxetine group
Drug: placebo pill — placebo pill orally 2 hours before the surgical procedure and at 24 hours after the surgical procedure
  Arms: placebo pill group

SUMMARY:
A total of 60 patients scheduled for thoracotomy with the aim of excision of pleural or lung cancer, will be randomized by the use of a computer-generated table of random numbers to receive duloxetine 60 mg orally 2 hours before the surgical procedure and at 24 hours after the surgical procedure or a placebo pill following the same time schedule.

ELIGIBILITY:
Inclusion criteria

* ASA I, II, and III patients scheduled for thoracotomy for pleural or lung cancer resection.
* Age above 18 years & less than 65 years.
* Adequate coagulation function within 30 days of surgery, defined as platelet count 100,000/mL or more, INR≤ 1.5, and partial thromboplastin time ≤40 seconds.

Exclusion criteria:

* Allergy to duloxetine or to local anesthetics.
* Patients with educational, psychiatric (untreated or poorly controlled schizophrenia, major depression, or bipolar disorder), or communication (language) barriers that would prevent understanding of the informed consent & preclude accurate assessment of postoperative pain and/or ability to answer questions about pain.
* Patients with severe renal and/or liver disease.
* History of chronic pain, long term narcotic use and/or antidepressants.
* Reasons for exclusion after randomization will be protocol violations or patient request.
* Fever, evidence of infection, or other coexisting medical conditions that would preclude epidural placement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Total dose of morphine needed to treat postoperative pain | 48 hours
  Total dose of morphine needed to treat postoperative pain over 48 hours of study period

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo University, Cairo, Egypt